CLINICAL TRIAL: NCT04307836
Title: A Prospective, Multicenter, No-treatment Controlled, Randomized, Open-label, Pivotal Study to Evaluate the Safety and Efficacy of DENEX, Renal Denervation Therapy, in Patients With Hypertension on no or 1-3 Antihypertensive Medications
Brief Title: DENEX, Renal Denervation Therapy, in Patients With Hypertension on no or 1-3 Antihypertensive Medications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kalos Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DN_P101
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-02

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases
Keywords: Hypertension; Renal Denervation; Uncontrolled hypertension
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DENEX Renal denervation (Experimental): Subjects are treated with the renal denervation procedure after randomization and maintained baseline anti-hypertensive medications
  Interventions: Device: Renal Denervation
- Control group (No Intervention): Subjects are not treated with the renal denervation, not sham, after randomization and maintained baseline anti-hypertensive medications

INTERVENTIONS:
Device: Renal Denervation — Renal Denervation: DENEX system
  Arms: DENEX Renal denervation

SUMMARY:
The objective of this study is to show that the safety and efficacy of renal denervation using DENEX, are superior to those of control group for the patients with hypertension on no or 1 to 3 antihypertensive medications.

DETAILED DESCRIPTION:
DENEX system developed by Handok Kalos Medical Inc. is a renal denervation system to efficiently block the sympathetic nerve of the kidney with minimal invasive procedure. It was developed to block the sympathetic nerves distributed in blood vessel wall by delivering high frequency energy to the renal artery for the purpose of treating hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 19 to 75 years old
* Subject should maintain the 0 to 3 antihypertensive medications of different classes, ACE-I, ARB, beta blocker, CCB or diuretics, without change for at least 4 weeks of run-in period between primary screening and secondary screening and for at least 3 months after the procedure
* Subject with 140 mmHg ≤ average office SBP < 180 mmHg and 90 mmHg ≤ office DBP < 120 mmHg at primary and secondary screening
* Subject with 135 mmHg ≤ average daytime ambulatory SBP <170 mmHg and 85 mmHg ≤ average daytime ambulatory DBP < 105 mmHg at secondary screening after the run-in period for at least 4 weeks

Exclusion Criteria:

* Subject with the anatomical findings in kidney or renal artery which preclude renal denervation
* Subject with type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus
* Subject with eGFR less than 40mL/min/1.73㎡
* Subject with a brachial circumference greater than 42 cm.
* Subject with secondary hypertension (except for sleep apnea patients)
* Subject with a medical history of cerebrovascular disease or severe cardiovascular disease within 12 months prior to obtaining the consent or patients newly diagnosed with such diseases before enrollment.
* Subject rehospitalized two or more times for hypertensive crisis within 12 months prior to obtaining consent or hospitalized for hypertensive crisis within three months prior to obtaining consent.
* Subject with chronic oxygen therapy or mechanical ventilation (except for sleep apnea)
* Subject with primary pulmonary hypertension

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2024-04-17 (Estimated)

PRIMARY OUTCOMES:
Changes in average daytime ambulatory systolic blood pressure at 3 months | from baseline at 3 months after the procedure
  Changes in average daytime ambulatory systolic blood pressure from baseline at 3 months after the procedure

SECONDARY OUTCOMES:
Changes in average 24hr ambulatory systolic blood pressure and diastolic blood pressure at 3, 6 and 12 months | from baseline at 3, 6 and 12 months after the procedure
  Changes in average 24hr ambulatory systolic blood pressure and diastolic blood pressure from baseline at 3, 6 and 12 months after the procedure
Changes in average office systolic blood pressure and diastolic blood pressure at 1, 3, 6 and 12 months | from baseline at 1, 3, 6 and 12 months after the procedure
  Changes in average office systolic blood pressure and diastolic blood pressure from baseline at 1,3, 6 and 12 months after the procedure
Changes in average daytime and nighttime ambulatory systolic blood pressure and diastolic blood pressure at 3, 6 and 12 months | from baseline at 3, 6 and 12 months after the procedure
  Changes in average daytime and nighttime ambulatory systolic blood pressure and diastolic blood pressure from baseline at 3, 6 and 12 months after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ki Yuk Chang, MD, Ph.D, Principal Investigator — Seoul St. Mary's Hospital
Locations (30):
- South Korea (30):
  - Bucheon St.Mary's Hospital, Bucheon-si
  - Hyewon Medical Foundation Sejong General Hospital, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Inje University Ilsan Paik Hospital, Ilsan
  - Gachon University Gil Medical Center, Incheon
  - Incheon St.Mary's Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Chonnam National University Hospital, Kwangju
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Yeouido St.Mary's Hospital, Seoul
  - St. Carollo Hospital, Suncheon
  - St. Vincent's Hospital, Suwon
  - Uijeongbu St.Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No